CLINICAL TRIAL: NCT04043975
Title: Japanese Prospective Real World Registry of Nivolumab Plus Ipilimumab in Subjects With Previously Untreated, Advanced or Metastatic Renal Cell Carcinoma (ARCC) Categorized Into IMDC Intermediate/Poor Risks (J-ENCORE)
Brief Title: A Study of Nivolumab Plus Ipilimumab in Participants With Renal Cell Cancer in the Real World Setting in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7CR
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Advanced or Metastatic Renal Cell Carcinoma
Keywords: Japanese; Observational Study
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with advanced or metastatic renal cell carcinoma (aRCC) receiving the combination of nivolumab plus ipilimumab as the first line of systemic therapy

SUMMARY:
The purpose of the observational study is to evaluate the safety and effectiveness of combination therapy with nivolumab and ipilimumab in Japanese participants with advanced or metastatic renal cell carcinoma (aRCC) in the real-world setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of Renal Cell Carcinoma (RCC)
* No prior systemic therapy for RCC
* Participants who are planned to start treatment with nivolumab and ipilimumab regimen in the timeframe between after IRB approval to enrollment-end date
* International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) risk category Intermediate/Poor

Exclusion Criteria:

* Participants who are enrolled in a post marketing safety study on nivolumab plus ipilimumab combination therapy in Japan
* Pregnant and/or lactating women
* Participants who are judged to be inappropriate by investigator

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of Japanese participants who will be treated with the combination of nivolumab+ipilimumab as first line of systematic therapy in the real world setting.
Sampling Method: Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of starting nivolumab plus ipilimumab to the date of death from any cause. (Up to 5 years)
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by Investigator | From date of starting nivolumab plus ipilimumab to the first date of documented progression, as determined by the investigators (as per RECIST 1.1 criteria), or death due to any cause, whichever occurs first. (Up to 5 years)
Change in tumor response over time | Up to 5 years
Duration of Response (DOR) | From first documentation of tumor response after the date of starting nivolumab plus ipilimumab to disease progression or death due to any cause, whichever occurs first. (Up to 5 years)
The quality of life by National Comprehensive Cancer Network/ Functional Assessment of Cancer Therapy (FACT)-Kidney Symptom Index 19 (NCCN-FACT FKSI-19) v2.0 | Up to 6 months
Number of participants with Adverse Events (AEs) | During the observation period or until 100 days after discontinuation of dosing with nivolumab and ipilimumab (Up to 5 years)
ORR on subsequent therapy | From initiation of a second line of therapy after discontinuation of first line nivolumab+ipilimumab treatment (Up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Tokyo, Japan

REFERENCES:
- [Derived] Sazuka T, Tatsugami K, Shirotake S, Hamamoto S, Nozawa M, Numakura K, Mizokami A, Kondo T, Naito S, Abe T, Ohba K, Kimura G, Onodera S, Yamaguchi K, Uemura H. Outcomes of Nivolumab-Plus-Ipilimumab in Metastatic Renal Cell Carcinoma: Second Interim Analysis of the J-ENCORE Study. Int J Urol. 2026 Jan;33(1):e70281. doi: 10.1111/iju.70281. Epub 2025 Nov 25. PMID 41292059
- [Derived] Nishimoto K, Kimura G, Sazuka T, Hamamoto S, Nozawa M, Numakura K, Mizokami A, Kondo T, Naito S, Abe T, Ohba K, Nagata M, Onodera S, Ito H, Uemura H. The Effectiveness and Safety Profile of Nivolumab-Plus-Ipilimumab in Previously Untreated Japanese Patients With Advanced or Metastatic Renal Cell Carcinoma (J-ENCORE Study). Int J Urol. 2025 Aug;32(8):961-972. doi: 10.1111/iju.70076. Epub 2025 Apr 24. PMID 40271863
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome